CLINICAL TRIAL: NCT04093492
Title: Preemie Prep For Parents (P3) Outpatient Mobile Intervention: Home Antenatal Prematurity Education
Brief Title: Preemie Prep For Parents (P3): Home Antenatal Prematurity Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mir A Basir, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00033902; R21HD092664 (NIH)
Record Dates: First submitted 2019-09-13; First posted 2019-09-18 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Premature Birth; Decision Making; Prenatal Care; Resuscitation; Infant, Premature
Keywords: gestational age; multi-media; mobile application; anxiety; clinical trial; random allocation
MeSH Terms: conditions — Premature Birth; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preemie Prep for Parents (P3) Outpatient Mobile Intervention (Experimental): The P3 mobile intervention in its current form sends participants text messages according to a schedule based on their gestational age. These text messages contain links to short videos uploaded to the P3 site, focusing on topics related to preterm labor and premature infants.
  Interventions: Other: Preemie Prep for Parents (P3) Outpatient Mobile Intervention
- ACOG links (Active Comparator): Participants in the active control condition will receive links to patient education handouts about preterm birth provided by the American College of Obstetricians and Gynecologists.
  Interventions: Other: ACOG links

INTERVENTIONS:
Other: Preemie Prep for Parents (P3) Outpatient Mobile Intervention — The P3 mobile intervention sends participants text messages according to a schedule based on their gestational age. These text messages contain links to short videos uploaded to the P3 site, focusing on topics related to preterm labor and premature infants.
  Arms: Preemie Prep for Parents (P3) Outpatient Mobile Intervention
Other: ACOG links — Participants in the active control condition will receive links to patient education handouts about preterm birth provided by the American College of Obstetricians and Gynecologists.
  Arms: ACOG links

SUMMARY:
The Preemie Prep for Parents (P3) mobile intervention will be tested in an outpatient population of pregnant women at risk of preterm birth and their partners. The study is a randomized controlled trial (RCT) comparing knowledge and preparedness for decision making between a group receiving the P3 texts and videos and a group receiving links to American College of Obstetricians and Gynecologists (ACOG) prematurity patient education handouts.

DETAILED DESCRIPTION:
This is a randomized controlled study focused on an outpatient population of pregnant women at risk of preterm birth and their partners. The objective is to test the efficacy of the Preemie Prep for Parents (P3) intervention on prematurity knowledge and preparedness for decision making.

Participants are recruited from their obstetric clinic appointment between weeks 16 and 21, and randomized 1:1 to either the P3 intervention, or access to electronic ACOG handouts (active control). Any participating partners are assigned to the same arm as their pregnant partner. The participants in the P3 group will then receive a schedule of automated text messages, with video links, up to twice a day. These videos and messages are based on information relevant to their gestational age.

At study entry, participants will complete measures of their health literacy, anxiety, decision self-efficacy, and subjective global health. As pregnancy continues, questionnaires will be sent to participants at the start of their 25th, 30th, and 34th weeks. These questionnaires will include Prematurity Knowledge Questionnaires (specific to their gestational age), a Preparation for Decision Making scale, and an anxiety measure. At study completion, within two weeks of either preterm childbirth or completion of the 34 week questionnaire, participants will be asked to also complete the Educational-Aid Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman or her partner
* At risk for preterm birth, as indicated by: history of spontaneous preterm birth (during the 34th week or earlier), shortened cervical length, multiple gestation, fetal growth restriction, chronic hypertension, history of preeclampsia, and/or diabetes requiring medications.
* Gestational age of 16-21 weeks at recruitment.
* Owns a smartphone.
* Able to speak English

Exclusion Criteria:

• Pregnancies with known significant birth defects.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Gender is a de facto criteria of inclusion, in that we will first be recruiting pregnant women. However, her partner or support person, should they wish to participate, may be of any gender.
Enrollment: 175 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Basir MA, McDonnell SM, Brazauskas R, Kim UO, Ahamed SI, McIntosh JJ, Pizur-Barnekow K, Pitt MB, Kruper A, Leuthner SR, Flynn KE. Effect of fathers in Preemie Prep for Parents (P3) program on couple's preterm birth preparedness. Patient Educ Couns. 2025 Mar;132:108599. doi: 10.1016/j.pec.2024.108599. Epub 2024 Dec 4. PMID 39647248
- [Derived] McDonnell SM, Flynn KE, McIntosh JJ, Brazauskas R, Kim UO, Ahamed SI, Basir MA. Video Education in Early Pregnancy and Parent Knowledge of Neonatal Resuscitation Options: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2344645. doi: 10.1001/jamanetworkopen.2023.44645. PMID 38010656
- [Derived] Flynn KE, McDonnell SM, Brazauskas R, Ahamed SI, McIntosh JJ, Pitt MB, Pizur-Barnekow K, Kim UO, Kruper A, Leuthner SR, Basir MA. Smartphone-Based Video Antenatal Preterm Birth Education: The Preemie Prep for Parents Randomized Clinical Trial. JAMA Pediatr. 2023 Jul 31;177(9):921-9. doi: 10.1001/jamapediatrics.2023.1586. Online ahead of print. PMID 37523163

RESULTS

PARTICIPANT FLOW:
Groups:
- Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Patients; Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons: The P3 mobile intervention in its current form sends participants text messages according to a schedule based on their gestational age. These text messages contain links to short videos uploaded to the P3 site, focusing on topics related to preterm labor and premature infants.
  Preemie Prep for Parents (P3) Outpatient Mobile Intervention: The P3 mobile intervention sends participants text messages according to a schedule based on their gestational age. These text messages contain links to short videos uploaded to the P3 site, focusing on topics related to preterm labor and premature infants.
- American College of Obstetricians and Gynecologists (ACOG) Links - Patients; American College of Obstetricians and Gynecologists (ACOG) Links - Support Persons: Participants in the active control condition will receive links to patient education handouts about preterm birth provided by the American College of Obstetricians and Gynecologists.
  ACOG links: Participants in the active control condition will receive links to patient education handouts about preterm birth provided by the American College of Obstetricians and Gynecologists.
Period: 25 Weeks Gestational Age (GA)
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Patients | American College of Obstetricians and Gynecologists (ACOG) Links - Patients | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | American College of Obstetricians and Gynecologists (ACOG) Links - Support Persons
Started | 60 | 60 | 34 | 21
Completed | 54 | 53 | 29 | 18
Not Completed | 6 | 7 | 5 | 3
Not completed — Delivered before assessment | 1 | 2 | 0 | 0
Not completed — No response | 5 | 5 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: 30 Weeks GA
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Patients | American College of Obstetricians and Gynecologists (ACOG) Links - Patients | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | American College of Obstetricians and Gynecologists (ACOG) Links - Support Persons
Started | 60 (Unless a participant chose to withdraw, they were considered enrolled and eligible for future assessments (i.e., a participant may have not responded to the 25 week questionnaire but still have been eligible and responded to the 30 week questionnaire). Therefore the number of participants who start a period may not be equal to the number who completed the previous period.) | 60 (Unless a participant chose to withdraw, they were considered enrolled and eligible for future assessments (i.e., a participant may have not responded to the 25 week questionnaire but still have been eligible and responded to the 30 week questionnaire). Therefore the number of participants who start a period may not be equal to the number who completed the previous period.) | 34 | 20
Completed | 52 | 52 | 29 | 18
Not Completed | 8 | 8 | 5 | 2
Not completed — Delivered before assessment | 1 | 2 | 0 | 0
Not completed — No response | 7 | 5 | 5 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: 34 Weeks GA
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Patients | American College of Obstetricians and Gynecologists (ACOG) Links - Patients | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | American College of Obstetricians and Gynecologists (ACOG) Links - Support Persons
Started | 60 (Unless a participant chose to withdraw, they were considered enrolled and eligible for future assessments (i.e., a participant may have not responded to the 25 week questionnaire but still have been eligible and responded to the 34 week questionnaire). Therefore the number of participants who start a period may not be equal to the number who completed the previous period.) | 60 (Unless a participant chose to withdraw, they were considered enrolled and eligible for future assessments (i.e., a participant may have not responded to the 25 week questionnaire but still have been eligible and responded to the 34 week questionnaire). Therefore the number of participants who start a period may not be equal to the number who completed the previous period.) | 34 | 20
Completed | 54 | 49 | 29 | 17
Not Completed | 6 | 11 | 5 | 3
Not completed — Delivered before assessment | 6 | 3 | 0 | 0
Not completed — No response | 0 | 7 | 5 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants; Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons: The P3 mobile intervention in its current form sends participants text messages according to a schedule based on their gestational age. These text messages contain links to short videos uploaded to the P3 site, focusing on topics related to preterm labor and premature infants.
  Preemie Prep for Parents (P3) Outpatient Mobile Intervention: The P3 mobile intervention sends participants text messages according to a schedule based on their gestational age. These text messages contain links to short videos uploaded to the P3 site, focusing on topics related to preterm labor and premature infants.
- ACOG Links - Pregnant Participants; ACOG Links - Support Persons: Participants in the active control condition will receive links to patient education handouts about preterm birth provided by the American College of Obstetricians and Gynecologists.
  ACOG links: Participants in the active control condition will receive links to patient education handouts about preterm birth provided by the American College of Obstetricians and Gynecologists.
- Total: Total of all reporting groups
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons | Total
Number analyzed (Participants) | 60 | 60 | 34 | 21 | 175
Age, Customized [Count of Participants; unit: Participants]
  20-24 years | 5 | 5 | 2 | 1 | 13
  25-34 years | 38 | 36 | 13 | 9 | 96
  35-46 | 17 | 19 | 17 | 11 | 64
  Missing | 0 | 0 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 1 | 2 | 123
  Male | 0 | 0 | 33 | 19 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Row population is divided by ethnicity (Hispanic/non-Hispanic).
  Participants
    non-Hispanic: number analyzed (Participants) | 57 | 53 | 28 | 20 | 158
    non-Hispanic: White | 40 | 37 | 21 | 15 | 113
    non-Hispanic: Black | 12 | 12 | 3 | 2 | 29
    non-Hispanic: American Indian | 0 | 0 | 0 | 0 | 0
    non-Hispanic: Asian | 1 | 3 | 1 | 0 | 5
    non-Hispanic: Native Hawaiian | 0 | 0 | 0 | 0 | 0
    non-Hispanic: More than one race | 4 | 1 | 2 | 3 | 10
    non-Hispanic: Missing | 0 | 0 | 1 | 0 | 1
    Hispanic: number analyzed (Participants) | 3 | 7 | 6 | 1 | 17
    Hispanic: White | 3 | 4 | 5 | 0 | 12
    Hispanic: Black | 0 | 2 | 0 | 0 | 2
    Hispanic: American Indian | 0 | 0 | 0 | 0 | 0
    Hispanic: Asian | 0 | 1 | 0 | 1 | 2
    Hispanic: Native Hawaiian | 0 | 0 | 0 | 0 | 0
    Hispanic: More than one race | 0 | 0 | 0 | 0 | 0
    Hispanic: Missing | 0 | 0 | 1 | 0 | 1
Gestational age at enrollment [Count of Participants; unit: Participants]
  16 weeks GA | 5 | 3 | 3 | 1 | 12
  17 weeks GA | 18 | 18 | 9 | 7 | 52
  18 weeks GA | 8 | 10 | 6 | 3 | 27
  19 weeks GA | 3 | 3 | 0 | 1 | 7
  20 weeks GA | 15 | 12 | 12 | 4 | 43
  21 weeks GA | 9 | 11 | 3 | 4 | 27
  22 weeks GA | 2 | 3 | 1 | 1 | 7
Education [Count of Participants; unit: Participants]
  9-12th grade, no diploma | 0 | 2 | 0 | 0 | 2
  High school diploma or equivalent | 8 | 10 | 4 | 3 | 25
  Some college | 13 | 9 | 11 | 3 | 36
  2-year degree | 7 | 8 | 5 | 1 | 21
  4-year degree | 17 | 16 | 11 | 6 | 50
  Graduate or professional degree | 15 | 15 | 3 | 8 | 41

OUTCOME MEASURES:

1. Primary Outcome: Parent Prematurity Knowledge Questionnaire
Description: Knowledge questionnaire developed by research team and tested through cognitive interviews, testing parental prematurity knowledge recommended by Eunice Kennedy Shriver National Institute of Child Health and Human Development. Subscales consist of long-term outcomes, variability in due date estimation, general prematurity knowledge, lowest gestational age needed for survival, factors influencing preterm birth outcome, treatment options, short-term outcomes, and advocacy. Subscale scores are summed to create a composite score. Versions of the questionnaire are slightly different at follow up points to ensure gestational age specific clinical relevance; the version at 25 weeks the questionnaire has 38 items. Therefore the range of scores is from 0-38, with higher scores indicating greater knowledge.
Time Frame: Assessed at participant's 25th week of pregnancy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 54 | 53 | 29 | 19
score on a scale | 30.3 (5.7) | 22.8 (5.9) | 29.3 (7.1) | 25.6 (4.1)

2. Primary Outcome: Parent Prematurity Knowledge Questionnaire
Description: Knowledge questionnaire developed by research team and tested through cognitive interviews, testing parental prematurity knowledge recommended by Eunice Kennedy Shriver National Institute of Child Health and Human Development. Subscales consist of long-term outcomes, variability in due date estimation, general prematurity knowledge, lowest gestational age needed for survival, factors influencing preterm birth outcome, treatment options, short-term outcomes, and advocacy. Subscale scores are summed to create a composite score. Versions of the questionnaire are slightly different at follow up points to ensure gestational age specific clinical relevance; the version at 30 weeks the questionnaire has 35 items. Therefore the range of scores is from 0-35, with higher scores indicating greater knowledge.
Time Frame: Assessed at participant's 30th week of pregnancy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 52 | 52 | 29 | 19
score on a scale | 29.2 (3.6) | 23.9 (5.1) | 27.9 (4.6) | 25.7 (3.5)

3. Primary Outcome: Parent Prematurity Knowledge Questionnaire
Description: Knowledge questionnaire developed by research team and tested through cognitive interviews, testing parental prematurity knowledge recommended by Eunice Kennedy Shriver National Institute of Child Health and Human Development. Subscales consist of long-term outcomes, variability in due date estimation, general prematurity knowledge, lowest gestational age needed for survival, factors influencing preterm birth outcome, treatment options, short-term outcomes, and advocacy. Subscale scores are summed to create a composite score. Versions of the questionnaire are slightly different at follow up points to ensure gestational age specific clinical relevance; the version at 34 weeks the questionnaire has 30 items. Therefore the range of scores is from 0-30, with higher scores indicating greater knowledge.
Time Frame: Assessed at participant's 34th week of pregnancy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 54 | 49 | 29 | 17
score on a scale | 25.8 (3.5) | 21.3 (4.8) | 24.2 (3.4) | 20.5 (6.3)

4. Primary Outcome: Preparation for Decision Making Scale
Description: Preparation for Decision Making Scale (Graham, O'Connor 1996, revised 2005). Scale ranges from a score of 10 to 50; these scores are converted to a 0-100 scale for ease of interpretation as recommended by the creators. Higher scores indicate higher perceived level of preparation for discussing a healthcare related decision.
Time Frame: Assessed at participant's 25th week of pregnancy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 54 | 53 | 28 | 19
score on a scale | 76.0 (18.3) | 52.3 (29.5) | 76.8 (16.3) | 57.1 (31.2)

5. Primary Outcome: Preparation for Decision Making Scale
Description: as for outcome 4
Time Frame: Assessed at participant's 30th week of pregnancy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 52 | 52 | 29 | 18
score on a scale | 76.3 (24.8) | 54.4 (25.1) | 69.2 (23.6) | 61.1 (14.9)

6. Primary Outcome: Preparation for Decision Making Scale
Description: as for outcome 4
Time Frame: Assessed at participant's 34th week of pregnancy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 54 | 49 | 29 | 16
score on a scale | 68.9 (25.1) | 54.2 (28.5) | 69.3 (24.0) | 63.6 (23.7)

7. Secondary Outcome: Anxiety
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Computerized Adaptive Test (CAT). As a Computer Adaptive Test (CAT), not all participants receive the same number of questions, but may range between 4 and 12 questions. The number and selection of questions is dependent on the previous responses. An average US adult has a score of 50 with a standard deviation of 10; the higher that t-score, the greater amount of anxiety the respondent is reporting.
Time Frame: Assessed at baseline
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participant; Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons: The P3 mobile intervention in its current form sends participants text messages according to a schedule based on their gestational age. These text messages contain links to short videos uploaded to the P3 site, focusing on topics related to preterm labor and premature infants.
  Preemie Prep for Parents (P3) Outpatient Mobile Intervention: The P3 mobile intervention sends participants text messages according to a schedule based on their gestational age. These text messages contain links to short videos uploaded to the P3 site, focusing on topics related to preterm labor and premature infants.
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participant | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 60 | 60 | 33 | 21
T-score | 53.7 (7.8) | 54.6 (8.2) | 49.9 (5.6) | 52.3 (8.7)

8. Secondary Outcome: Anxiety
Description: as for outcome 7
Time Frame: Assessed at participant's 25th week of pregnancy.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 54 | 53 | 29 | 19
T-score | 53.6 (7.9) | 53.8 (8.2) | 49.5 (7.2) | 52.4 (6.4)

9. Secondary Outcome: Anxiety
Description: as for outcome 7
Time Frame: Assessed at participant's 30th week of pregnancy.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 52 | 52 | 29 | 20
T-score | 52.7 (7.7) | 55.3 (6.8) | 48.5 (7.9) | 53.0 (8.6)

10. Secondary Outcome: Anxiety
Description: as for outcome 7
Time Frame: Assessed at participant's 34th week of pregnancy.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 54 | 49 | 29 | 16
T-score | 53.5 (9.2) | 55.5 (8.2) | 50.9 (9.0) | 53.0 (7.2)

11. Secondary Outcome: Decision Self-Efficacy
Description: Decision Self-Efficacy Scale (O'Connor, 1995). Scale ranges from a score of 0 to 44; these scores are converted to a 0-100 scale for ease of interpretation as recommended by the creators. Higher scores indicate higher perceived level of decision self-efficacy.
Time Frame: Assessed at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 60 | 60 | 38 | 16
score on a scale | 92.1 (11.3) | 91.6 (10.3) | 88.3 (13.4) | 95.0 (8.2)

12. Secondary Outcome: Decision Self-Efficacy
Description: as for outcome 11
Time Frame: Assessed at 34 weeks of pregnancy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Pregnant Participants | ACOG Links - Pregnant Participants | Preemie Prep for Parents (P3) Outpatient Mobile Intervention - Support Persons | ACOG Links - Support Persons
Number analyzed (Participants) | 54 | 49 | 29 | 16
score on a scale | 89.3 (12.1) | 85.8 (17.6) | 86.8 (12.3) | 86.8 (15.2)

ADVERSE EVENTS:
Time Frame: Duration of study participation; total weeks depends on gestational age at enrollment (16 to 21 weeks GA) and gestational age at delivery (i.e., up to 27 weeks).
Description: Adverse events were not assessed for support persons, as we did not have access to their medical records.
Arm/Group | Preemie Prep for Parents (P3) Outpatient Mobile Intervention | ACOG Links
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT04093492/Prot_SAP_000.pdf